CLINICAL TRIAL: NCT04107467
Title: Mechanical Ventilation Epidemiology in Argentina. EpVAr Multicenter Study.
Brief Title: Mechanical Ventilation Epidemiology in Argentina.
Acronym: EpVAr2019
Status: Completed | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Physical and Respiratory Therapist, Head of Physical and Respiratory Therapist Department, Sanatorio Anchorena, Buenos Aires, Argentina, Argentinian Intensive Care Society
Other Study IDs: EpVAr
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Respiration, Artificial; Epidemiology
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
How is the epidemiology of mechanically ventilated patients in the intensive care units of Argentina?

DETAILED DESCRIPTION:
Mechanical ventilation is an indispensable tool in life support and one of the interventions that characterizes intensive care units (ICU).

Epidemiological studies have allowed us to improve knowledge and optimize the treatment of patients with acute respiratory failure.

In Latin America the epidemiological data of mechanical ventilation is poor.

Primary goal of this national, observational, prospective, multicentric epidemiological study: to analyze the survival and describe epidemiological features of patients receiving mechanical ventilation in the Intensive Care Units of Argentina.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients requiring Mechanical Ventilation at least for 12 hours
* ICU patients who initiate Mechanical Ventilation in the Operation Room or the Emergency Room
* ICU patients who initiate Mechanical Ventilation in other institution.

Exclusion Criteria:

* Patients under 18 years old
* Patients in Pediatric ICU
* Patients in Coronary ICU
* Patients without requirements of Mechanical Ventilation
* Patients who have been discharged from ICU and re-enter during the enrollment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who require mechanical ventilation for at least 12 hours in the argentinians ICU will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Survival in the ICU | Up to 28 days after the enrollment
  "Survival in the ICU" will be measured as YES or NO at day 28 after the enrollment.

SECONDARY OUTCOMES:
Main reason of Invasive Mechanical Ventilation | 1 day
  1. Acute respiratory failure in patient with chronic respiratory failure: A)Chronic Obstructive Pulmonary Disease, B) Asthma, C) Other Chronic Obstructive Pulmonary Disease (Idiopathic pulmonary fibrosis, Cystic Fibrosis, Interstitial disease).
  2. Acute Respiratory Failure: A) Acute Respiratory Distress Syndrome, B) Postoperative, C) Acute Heart Failure, D) Aspiration, E) Pneumonia, F) Sepsis, G) Trauma, H) Cardiac arrest, I)Others.
  3. Coma: A)Metabolic, B)Overdose, Intoxication, C)Stroke, D)Brain trauma.
  4. Neuromuscular disease
Ventilatory Modes and setting | Up to 10 days
  Volume Control Ventilation, Pressure Control Ventilation, Pressure Support Ventilation, Synchronized Intermittent Mandatory Ventilation, Other (Proportional Assist Ventilation, Neurally Adjusted Ventilation, Airway Pressure Release Ventilation)
Tidal Volume | Up to 10 days
  Set tidal volume in mililiters
Weaning and mortality | Up to 28 days
  Weaning characteristics and outcome of the patient in terms of mortality.
Noninvasive ventilation during weaning and mortality | Up to 28 days
  The use of NIV during weaning and the outcome of the patient in terms of mortality
Incidence of delirium | Up to 28 days
  Delirium measured with the CAM- ICU.
Incidence of ICU acquired weakness | Up to 28 days
  Periphereal muscle weakness measured with MRC defined as a total value of less than 48 points.
Incidence of tracheostomy | Up to 28 days
  Presence of tracheostomy
Sedation and analgesia in mechanical ventilation | Up to 28 days
  Implementation of sedation and analgesia during the period of mechanical ventilation.
Peak Pressure | Up to 10 days
  Monitored Peak Pressure in centimeters of water
Plateau Pressure | Up to 10 days
  Monitored Plateau Pressure in centimeters of water
Applied PEEP | Up to 10 days
  Set PEEP in centimeters of water
Total PEEP | Up to 10 days
  Monitored total PEEP in centimeters of water
Driving Pressure | Up to 10 days
  Monitored Driving Pressure in centimeters of water as the difference between Total PEEP and Plateau Pressure in centimeters of water

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Plotnikow, RT, Principal Investigator — Sanatorio Anchorena
Locations (154):
- Argentina (154):
  - Hospital Fiorito, Avellaneda
  - Sanatorio Norte SRL, Avellaneda
  - Hospital Italiano Regional del Sur, Bahía Blanca
  - Hospital privado Dr Raul Matera, Bahía Blanca
  - Hospital Area Programa Bariloche "Ramón Carrillo", Bariloche
  - Cemic H.U. Pombo, Buenos Aires
  - CEMIC H.U. Saavedra, Buenos Aires
  - Clinica La Sagrada Familia, Buenos Aires
  - Clinica y Maternidad Suizo Argentina, Buenos Aires
  - Clinica Zabala, Buenos Aires
  - Clínica Adventista Belgrano, Buenos Aires
  - Clínica Bazterrica, Buenos Aires
  - Clínica Pasteleros, Buenos Aires
  - Complejo Medico de la Policia Federal Churruca Visca, Buenos Aires
  - Cínica de los Virreyes, Buenos Aires
  - Hospital Alemán, Buenos Aires
  - Hospital Alvarez, Buenos Aires
  - Hospital de Clínicas José de San Martín, Buenos Aires
  - Hospital de Rehabilitación Respiratoria María Ferrer, Buenos Aires
  - Hospital de Trauma y Emergencia Dr. Federico Abete, Buenos Aires
  - Hospital Dr D. Velez Sarsfield, Buenos Aires
  - Hospital Fernandez, Buenos Aires
  - Hospital Francisco Javier Muñiz, Buenos Aires
  - Hospital Generall de Agudos Dr Cosme Argerich, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Naval Pedro Mallo, Buenos Aires
  - Hospital Piñero, Buenos Aires
  - Hospital Ramos Mejía, Buenos Aires
  - Hospital Santojanni SRS, Buenos Aires
  - Hospital Santojanni, Buenos Aires
  - Hospital Sirio Libanes, Buenos Aires
  - Hospital Universitario Fundación Favaloro-UTI 1, Buenos Aires
  - Hospital Universitario Fundación Favaloro-UTI 2, Buenos Aires
  - Hospital Universitario UAI, Buenos Aires
  - HZGA Dr alberto Balestrini, Buenos Aires
  - Instituto Argentino de Diagnostico y Tratamiento, Buenos Aires
  - Instituto de Trasplante y Alta Complejidad, Buenos Aires
  - Instituto Lanari, Buenos Aires
  - Instituto Médico de Alta Complejidad, Buenos Aires
  - Sanatorio Anchorena, Buenos Aires
  - Sanatorio Colegiales, Buenos Aires
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Sanatorio de la Trinidad Palermo, Buenos Aires
  - Sanatorio de los Arcos, Buenos Aires
  - Sanatorio Finochietto, Buenos Aires
  - Sanatorio Mater Dei, Buenos Aires
  - Sanatorio Otamendi, Buenos Aires
  - Htal de alta complejidad cuenca alta SAMIC, Cañuelas
  - Hospital Municipal de Agudos Dr. Pedro Ecay, Carmen de Patagones
  - Instituto Medico de la Comunidad, Catamarca
  - Hospital Municipal del Carmen de Chacabuco, Chacabuco
  - Hospital de Chivilcoy, Chivilcoy
  - Policlinico Modelo Cipolletti, Cipolletti
  - Hospital Carrillo de Ciudadela, Ciudadela
  - Clinica del Valle, Comodoro Rivadavia
  - Hospital Regional V Sanguinetti, Comodoro Rivadavia
  - Hospital Zonal Alvear, Comodoro Rivadavia
  - Hospital Justo José de Urquiza, Concepción del Uruguay
  - Hospital Escuela Gral José de San Martín, Corrientes
  - Instituto de Cardiologia Juana Francisca Cabral, Corrientes
  - Clinica Chutro, Córdoba
  - Clínica Santa Maria, Córdoba
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Hospital Córdoba, Córdoba
  - Hospital Italiano, Córdoba
  - Hospital Misericordia Nuevo Siglo, Córdoba
  - Hospital Municipal Principe de Asturias, Córdoba
  - Hospital Privado de Cordoba, Córdoba
  - Hospital Publico Provincial de la Ciudad de Córdoba, Córdoba
  - Hospital San Roque, Córdoba
  - Sanatorio Allende Cerro, Córdoba
  - Sanatorio Allende Nueva Córdoba, Córdoba
  - Sanatorio Privado del Intenterio SRL, Córdoba
  - Hospital Central de Formosa, Formosa
  - Sanatorio Juan XXIII, General Roca
  - Hospital Simplemente Evita, González Catán
  - Hospital Eva Peron, Granadero Baigorria
  - Hospital Profesor Dr Luis Guemes, Haedo
  - Clínica la pequeña Familia, Junín
  - Clínica Argentina, La Pampa
  - HIEA y C "San Juan de Dios", La Plata
  - HIGA San Martín de La Plata, La Plata
  - HIGA San Roque, La Plata
  - Hospital español, La Plata
  - Hospital Italiano de La Plata, La Plata
  - Instituto Médico Platense, La Plata
  - Ipensa, La Plata
  - Sanatorio Adventista del Plata, La Plata
  - HIGA Luisa Cravenna de Gandulfo, Lomas de Zamora
  - Clinica 25 de Mayo, Mar del Plata
  - HIGA Dr Oscar Alende, Mar del Plata
  - Clinica Santa Maria, Mendoza
  - Clinica Sociedad Española de Socorros Mutuos de Mendoza, Mendoza
  - Hospital Central, Mendoza
  - Hospital del Carmen, Mendoza
  - Hospital Luis C Lagomaggiore, Mendoza
  - Hospital Santa Isabel de Hungría, Mendoza
  - Hospital Eva Perón, Merlo
  - Clínica Monte Grande, Monte Grande
  - HZGA Mariano y Luciano de la Vega, Moreno
  - Hospital de Morón, Morón
  - Hospital Nacional A. Posadas, Morón
  - Sanatorio Clínica Modelo de Moron, Morón
  - Hospital Municipal Emilio Ferreyra, Necochea
  - Clinica CMIC, Neuquén
  - Clínica Pasteur, Neuquén
  - Clínica San Agustín, Neuquén
  - Clinica Olivos, Olivos
  - Hospital Militar Regional de Parana, Paraná
  - HIGA San Jose de Pergamino, Pergamino
  - Hospital Universitario Austral, Pilar
  - Hospital Municipal de Pinamar, Pinamar
  - Hospital Escuela de Agudos Dr. Ramon Madariaga, Posadas
  - Hospital Público Autogestión SAMIC el Dorado, Posadas
  - Hospital de Autogestión Samic Iguazú, Puerto Iguazú
  - Sanatorio de la Ciudad S.R.L, Puerto Madryn
  - Sanatorio de la Trinidad Quilmes, Quilmes
  - Sanatorio de la Trinidad Ramos Mejía, Ramos Mejía
  - Hospital central Reconquista, Reconquista
  - Hospital Dr. Julio Perrando, Resistencia
  - Hospital Español de Rosario, Rosario
  - Policlinico PAMI 1, Rosario
  - Sanatorio Mapaci, Rosario
  - Sanatorio Parque, Rosario
  - Hospital del Sr. del Milagro, Salta
  - Hospital Papa Francisco, Salta
  - Hospital Publico de Auogestión Dr Arturo Oñativia, Salta
  - HPGD San Bernardo, Salta
  - HIGA Petrona V. de Cordero de San Fernando, San Fernando
  - Sanatorio de la Trinidad San Isidro, San Isidro
  - Sanatorio Las Lomas, San Isidro
  - Centro de Cuidados Intensivos, San Juan
  - Clinica Santa Clara de la Porvincia de San Juan, San Juan
  - Hospital Dr Guillermo Rawson, San Juan
  - Hospital Público descentralizado Dr. Marcial Vicente Quiroga., San Juan
  - Hospital Italiano de San Justo, San Justo
  - Hospital Madre Catalina, San Luis
  - Hospital San Luis, San Luis
  - Hospital Centro de Salud Zenón Santillán, San Miguel de Tucumán
  - Hospital de clínica Presidente Doctor Nicolas Avellaneda, San Miguel de Tucumán
  - Sanatorio Lavalle, San Salvador de Jujuy
  - Sanatorio Nuestra Sra del Rosario, San Salvador de Jujuy
  - Htal Cullen de Santa Fe, Santa Fe
  - Sanatorio Español, Santa Fe
  - Sanatorio Santa Fe, Santa Fe
  - Sanatorio Santa Fé, Santa Fe
  - Centro Integral de Salud Banda, Santiago del Estero
  - Hospital regional Dr. Ramon Carrillo, Santiago del Estero
  - Hospital Ramón Santamarina, Tandil
  - Sanatorio Juncal, Temperley
  - Hospital Regional de Ushuaia, Ushuaia
  - Hospital Nodal Dr. Alejandro Gutierrez, Venado Tuerto
  - Hospital Houssay, Vicente López
  - Hospital Artemides Zatti, Viedma

REFERENCES:
- [Background] Protti A, Cressoni M, Santini A, Langer T, Mietto C, Febres D, Chierichetti M, Coppola S, Conte G, Gatti S, Leopardi O, Masson S, Lombardi L, Lazzerini M, Rampoldi E, Cadringher P, Gattinoni L. Lung stress and strain during mechanical ventilation: any safe threshold? Am J Respir Crit Care Med. 2011 May 15;183(10):1354-62. doi: 10.1164/rccm.201010-1757OC. Epub 2011 Feb 4. PMID 21297069
- [Background] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Esteban A, Frutos F, Tobin MJ, Alia I, Solsona JF, Valverdu I, Fernandez R, de la Cal MA, Benito S, Tomas R, et al. A comparison of four methods of weaning patients from mechanical ventilation. Spanish Lung Failure Collaborative Group. N Engl J Med. 1995 Feb 9;332(6):345-50. doi: 10.1056/NEJM199502093320601. PMID 7823995
- [Result] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224
- [Result] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Result] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Result] Azevedo LC, Park M, Salluh JI, Rea-Neto A, Souza-Dantas VC, Varaschin P, Oliveira MC, Tierno PF, dal-Pizzol F, Silva UV, Knibel M, Nassar AP Jr, Alves RA, Ferreira JC, Teixeira C, Rezende V, Martinez A, Luciano PM, Schettino G, Soares M; ERICC (Epidemiology of Respiratory Insufficiency in Critical Care) investigators. Clinical outcomes of patients requiring ventilatory support in Brazilian intensive care units: a multicenter, prospective, cohort study. Crit Care. 2013 Apr 4;17(2):R63. doi: 10.1186/cc12594. PMID 23557378
- [Result] Tomicic V, Espinoza M, Andresen M, Molina J, Calvo M, Ugarte H, Godoy J, Galvez S, Maurelia JC, Delgado I, Esteban A; Grupo Chileno para el Estudio de la Ventilacion Mecanica. [Characteristics and factors associated with mortality in patients receiving mechanical ventilation: first Chilean multicenter study]. Rev Med Chil. 2008 Aug;136(8):959-67. Epub 2008 Oct 7. Spanish. PMID 18949178
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Charlson ME, Charlson RE, Peterson JC, Marinopoulos SS, Briggs WM, Hollenberg JP. The Charlson comorbidity index is adapted to predict costs of chronic disease in primary care patients. J Clin Epidemiol. 2008 Dec;61(12):1234-1240. doi: 10.1016/j.jclinepi.2008.01.006. Epub 2008 Jul 10. PMID 18619805
- [Result] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Fabregas N, Ewig S, Torres A, El-Ebiary M, Ramirez J, de La Bellacasa JP, Bauer T, Cabello H. Clinical diagnosis of ventilator associated pneumonia revisited: comparative validation using immediate post-mortem lung biopsies. Thorax. 1999 Oct;54(10):867-73. doi: 10.1136/thx.54.10.867. PMID 10491448
- [Result] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Result] Chanques G, Jaber S, Barbotte E, Violet S, Sebbane M, Perrigault PF, Mann C, Lefrant JY, Eledjam JJ. Impact of systematic evaluation of pain and agitation in an intensive care unit. Crit Care Med. 2006 Jun;34(6):1691-9. doi: 10.1097/01.CCM.0000218416.62457.56. PMID 16625136
- [Result] Gelinas C, Johnston C. Pain assessment in the critically ill ventilated adult: validation of the Critical-Care Pain Observation Tool and physiologic indicators. Clin J Pain. 2007 Jul-Aug;23(6):497-505. doi: 10.1097/AJP.0b013e31806a23fb. PMID 17575489
- See also: Free software environment for statistical computing and graphics — http://www.r-project.org